CLINICAL TRIAL: NCT04768816
Title: Clinical Effect and Safety of Autologous Umbilical Cord Blood Transfusion in the Treatment of Autism Spectrum Disorder
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, Xiao Huimei, Dr, Guangdong Women and Children Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GuangdongWCHASD
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Safety Issues;Effect of Drugs
Keywords: Autism Spectrum Disorder;Autologous Umbilical Cord Blood;safety;effect
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): Placebo 0.9% sodium chloride infusion any time after entering the Placebo Group, doses is 20-30ml. The infusion speed is 1ml/min.
  Interventions: Drug: 0.9% Sodium Chloride
- Experimental (Experimental): Autologous Umbilical Cord Blood Mononuclear Cells Therapy any time after the diagnosis of cerebral palsy, doses is 20-30ml (total Mononuclear cells#1*10^7/kg). The infusion speed is 1ml/min.
  Interventions: Biological: Autologous Umbilical Cord Blood

INTERVENTIONS:
Drug: 0.9% Sodium Chloride — 0.9% Sodium Chloride in control group
  Arms: Placebo Comparator
Biological: Autologous Umbilical Cord Blood — Autologous Umbilical Cord Blood Mononuclear Cells Therapy in Autism Spectrum Disorder for safety and effect evaluation.
  Other Names: Autologous Umbilical Cord Blood Mononuclear Cells Therapy
  Arms: Experimental

SUMMARY:
To study the clinical efficacy and safety of autologous umbilical cord blood transfusion in the treatment of autism spectrum disorder.

DETAILED DESCRIPTION:
This is a Phase 1 clinical trial that constitutes two time points cohorts with participants who will receive intravenous autologous umbilical cord blood and 0.9% sodium chloride respectively. The timing of treatment is any time after the diagnosis of autism spectrum disorder. The investigator will proceed the groups during the same period.

1. Demographic Data and Baseline Characteristics of the Studied Group were collected:

   * Basic patient's information survey
   * Medical history
   * Physical examination
   * Basic blood test result
   * Autism Behavior Checklist,CARS before the treatment
   * Brain Magnetic Resonance Imaging-Diffusion Tensor Imaging (MRIDTI) before the treatment
   * Neurocognitive function test before the treatment
2. Assessment of clinical condition in the course by measurement of blood pressure, heart and respiratory rates, temperature and adverse events was recorded.
3. Autologous cord blood doses is 20-30ml (total Mononuclear cells# 1*10^7/kg)#the infusion speed is 1ml/min, and with same volume of 0.9% sodium chloride as placebo.
4. The follow-up: clinical test until 24th month in 3 month gaps.

ELIGIBILITY:
Inclusion Criteria:

* • A patient who was diagnosed with ASD.

Exclusion Criteria:

* • In case a patient underwent a surgical procedure, or was administered autologous cord blood within one year before participating in a clinical trial.

  * Accompanied by a serious disease, such as chromosome abnormality, etc.
  * In case where a patient's medical condition is judged to be maladapted by a researcher.
  * In case a patient or his or her legal representative doesn't agree to participation in a clinical trial.
  * A patient having a predisposition to allergies.
  * A patient having serious disorders in the liver, kidney, and cardiopulmonary function.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ABC | up to 24 months after therapy at a 3-month interval
  The Change of ABC score is used to assess the social and behavior function of the children who were diagnosised as ASD.
CARS | up to 24 months after therapy at a 3-month interval
  The Change of CARS score is used to assess the social and behavior function of the children who were diagnosised as ASD.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Women and Children's Hospital and Health Institute, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dawson G, Sun JM, Davlantis KS, Murias M, Franz L, Troy J, Simmons R, Sabatos-DeVito M, Durham R, Kurtzberg J. Autologous Cord Blood Infusions Are Safe and Feasible in Young Children with Autism Spectrum Disorder: Results of a Single-Center Phase I Open-Label Trial. Stem Cells Transl Med. 2017 May;6(5):1332-1339. doi: 10.1002/sctm.16-0474. Epub 2017 Apr 5. PMID 28378499
- [Background] Dawson G, Sun JM, Baker J, Carpenter K, Compton S, Deaver M, Franz L, Heilbron N, Herold B, Horrigan J, Howard J, Kosinski A, Major S, Murias M, Page K, Prasad VK, Sabatos-DeVito M, Sanfilippo F, Sikich L, Simmons R, Song A, Vermeer S, Waters-Pick B, Troy J, Kurtzberg J. A Phase II Randomized Clinical Trial of the Safety and Efficacy of Intravenous Umbilical Cord Blood Infusion for Treatment of Children with Autism Spectrum Disorder. J Pediatr. 2020 Jul;222:164-173.e5. doi: 10.1016/j.jpeds.2020.03.011. Epub 2020 May 19. PMID 32444220